CLINICAL TRIAL: NCT03164538
Title: A Psychological-behavioral Intervention to Increase Activity in Type 2 Diabetes: a 16-week Randomized Controlled Trial
Brief Title: A Psychological-behavioral Intervention to Increase Activity in Type 2 Diabetes
Acronym: BEHOLD-16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Chief of Psychiatry for Clinical Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001113
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology + Motivational Interviewing (Experimental): Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing
- Diabetes Education (Active Comparator): Participants will speak on the telephone each week with a study trainer. During these calls, the trainer will provide education about a health behavior related to diabetes health (physical activity, medication adherence, diet).
  Interventions: Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — Participants randomized to PP-MI will receive a treatment manual. For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. Following randomization, participants will engage in weekly, 30-minute phone calls over the next 16 weeks. Participants will independently complete PP exercises and MI-based goals between phone sessions and review them during phone sessions. PP and MI components will be delivered stepwise within sessions (rather than intertwined).
  Arms: Positive Psychology + Motivational Interviewing
Behavioral: Diabetes Education — Each week, participants will learn about a different health behavior topic related to diabetes health. As an attentional control, this condition has a parallel structure to the experimental arm with a treatment manual, weekly assignments, and weekly calls to review assignments.
  Arms: Diabetes Education

SUMMARY:
The focus of this study is to examine the feasibility, acceptability, and impact of a customized, combined positive psychology and motivational interviewing (PP-MI) health behavior intervention in a group of patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The investigators will compare a combined positive psychology and motivational interviewing (PP-MI) intervention that is adapted for patients with T2D to a diabetes education intervention (control) in a randomized controlled trial. The investigators will enroll 70 participants, who will be randomized to either a 16-week PP-MI health behavior intervention or an 16-week diabetes education intervention.

In this project, the investigators plan to do the following:

1. Examine the feasibility and acceptability of a 16-week, telephone-delivered health behavior intervention utilizing PP exercises and MI with systematic goal-setting.
2. Determine whether the PP-MI intervention leads to greater increases in physical activity than the education intervention in T2D patients.
3. Explore the impact of the PP-MI intervention on other psychological, behavioral, and medical outcomes, compared to the education intervention.

Participants will undergo an initial screening visit during which they will meet with study staff in person. At this visit, study eligibility will be confirmed, and eligible and willing participants will be enrolled. Following enrollment, participants will complete self-report measures, and vital signs and A1c will be measured. They then will take home and wear an accelerometer for one week, to measure baseline physical activity.

Baseline information about enrolled participants will be obtained from the participants, care providers, and the electronic medical record as required for characterization of the population. This information will include data regarding medical history (type 2 diabetes mellitus), current medical variables (conditions affecting physical activity), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will undergo a second in-person visit once adequate baseline physical activity data has been obtained. In this visit, accelerometer data will be reviewed to ensure that adequate baseline activity was captured. If so, participants will be randomized to either the PP-MI or diabetes education condition, then begin the study intervention. During this second in-person visit, participants will receive either a PP-MI or diabetes education treatment manual, depending on randomization.

For the PP-MI intervention:

For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. At subsequent sessions, participants will review the prior week's PP exercise and learn about a new exercise, then will review the prior week's physical activity goal and set a new one.

For the diabetes education intervention:

Each week, participants will learn about a different health behavior topic related to diabetes health. This includes information about diabetes self-monitoring, medication adherence, having a heart-healthy diet, and being physically active.

Participants will complete the remaining sessions by phone approximately weekly over the next 16 weeks. Phone sessions will last approximately 30 minutes, with PP-MI and physical activity assignments completed between phone sessions. PP and MI will be delivered step-wise within sessions (rather than intertwined) based on our experience, participant feedback, and pilot work. If a week is missed, the session will not be skipped, but rather the intervention will be completed sequentially (with participants who miss weeks then missing the final sessions), with the exception of the final visit, which skips to Planning for the Future in all cases.

Participants will undergo an in-person follow-up assessment at 16 weeks. At this session, participants will repeat self-report assessments that were administered at baseline. Vital signs and a blood sample will again be collected at this in-person visit. Prior to this assessment, participants will wear an accelerometer for 7 days to measure physical activity. Participants will also undergo a phone follow-up assessment at 24 weeks. During this session over the phone, participants will repeat self-report assessments that were administered at baseline. Finally, prior to this follow-up, participants will wear another accelerometer for 7 days to measure physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. T2D. Eligible patients will meet American Diabetes Association (ADA) criteria for T2D (e.g., HbA1c [A1C] ≥6.5%, fasting glucose ≥126 mg/d), with diagnosis confirmed by their diabetes clinician and/or medical record review.
2. Low physical activity. Low physical activity will be defined as ≤150 minutes/week of MVPA (corresponding to ADA recommendations for moderate or greater intensity aerobic physical activity). Physical activity will be measured using a brief questionnaire adapted from the International Physical Activity Questionnaire (IPAQ).

Exclusion Criteria:

1. Cognitive impairment precluding consent or meaningful participation.
2. Lack of phone availability.
3. Inability to read/write in English.
4. Additional medical conditions (e.g., severe arthritis) that preclude physical activity.
5. Enrollment in mind-body programs, lifestyle intervention programs (e.g., cardiac rehabilitation), or other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Psychology + Motivational Interviewing: Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Positive Psychology + Motivational Interviewing: Participants randomized to PP-MI will receive a treatment manual. For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. Following randomization, participants will engage in weekly, 30-minute phone calls over the next 16 weeks. Participants will independently complete PP exercises and MI-based goals between phone sessions and review them during phone sessions.
Period: Overall Study
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Started | 35 | 35
Completed | 28 | 29
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.2) | 62.9 (10.7) | 63.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 24 | 30 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Moderate-Vigorous Physical Activity [Mean (Standard Deviation); unit: minutes/day] — ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at Baseline, Week 16, and Week 24 to assess the feasibility of doing so and to ensure adequate capture of physical activity.
  minutes/day | 13.66 (13.15) | 13.67 (12.12) | 13.66 (12.55)
Physical Activity [Mean (Standard Deviation); unit: steps/day] — Measured by Actigraph accelerometer, in number of steps per day.
  steps/day | 4706 (2389) | 4805 (1993) | 4756 (2184)
Sedentary Time [Mean (Standard Deviation); unit: minutes/day] — Measured by Actigraph accelerometer, in minutes per day.
  minutes/day | 551.40 (98.74) | 499.66 (78.33) | 525.53 (92.23)
Positive Affect [Mean (Standard Deviation); unit: score on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
  score on a scale | 35.74 (6.87) | 33.51 (7.54) | 34.63 (7.25)
Optimism [Mean (Standard Deviation); unit: score on a scale] — Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism.
  score on a scale | 15.94 (5.64) | 17.20 (4.73) | 16.57 (5.20)
Self-Efficacy for Exercise [Mean (Standard Deviation); unit: score on a scale] — Measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assess self-efficacy barriers to exercise (Range: 0-90). Higher scores indicate higher efficacy expectations in relation to exercising.
  score on a scale | 50.06 (19.63) | 55.43 (21.66) | 52.74 (20.69)
Depression [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
  score on a scale | 3.63 (3.87) | 4.00 (3.61) | 3.81 (3.72)
Anxiety [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
  score on a scale | 5.37 (4.16) | 5.60 (4.31) | 5.49 (4.21)
Resilience [Mean (Standard Deviation); unit: score on a scale] — Measured by the Brief Resilience Scale (BRS), a reliable scale which assesses a person's ability to recover from stress despite adversity (Range: 6-30). Higher scores indicate more resilience.
  score on a scale | 17.86 (2.32) | 18.06 (1.63) | 17.96 (1.99)
Perceived Social Support (MSPSS) [Mean (Standard Deviation); unit: score on a scale] — Measured by the Multidimensional Scale of Perceived Social Support (MSPSS), a scale that measures subjectively reported social support (Range: 12-84). Higher scores indicate more subjectively reported social support.
  score on a scale | 64.06 (18.25) | 63.14 (18.25) | 63.60 (18.12)
Diabetes Self-Care [Mean (Standard Deviation); unit: score on a scale] — Measured by the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more diabetes self-care activities.
  score on a scale | 3.17 (1.02) | 2.27 (1.09) | 2.72 (1.14)
Medication Adherence [Mean (Standard Deviation); unit: percentage of medication taken] — Measured by Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum: 100. Higher scores indicate greater levels of medication adherence.
  percentage of medication taken | 91 (22) | 93 (14) | 92 (18)
Self-Reported Physical Activity [Mean (Standard Deviation); unit: MET minutes per week] — Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week.
  MET minutes per week | 633.82 (560.97) | 1914.87 (4374.98) | 1274.34 (3162.72)
Physical Function [Mean (Standard Deviation); unit: score on a scale] — Measured by the 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS), a well-validated measure of physical function that is highly responsive to changes in a patient's physical function status (Range: 20-100). Higher scores indicate better physical function.
  score on a scale | 92.77 (5.50) | 90.31 (10.92) | 91.54 (8.67)
Pain-Related Disability [Mean (Standard Deviation); unit: score on a scale] — Measured by the Pain Disability Index (PDI), a well-validated measure of the extent to which pain interferes with different daily activities (Range 0-70). Higher scores indicate greater interference from pain. Population: One participant did not complete this measure at baseline.
  score on a scale
    number analyzed (Participants) | 35 | 34 | 69
    (all) | 8.77 (10.36) | 13.71 (15.15) | 11.20 (13.09)
Weight [Mean (Standard Deviation); unit: pounds] | 195.10 (34.02) | 194.05 (40.85) | 194.57 (37.32)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.98 (4.47) | 31.08 (5.58) | 31.03 (5.02)
Blood Pressure (systolic) [Mean (Standard Deviation); unit: millimeters of mercury] | 139.63 (11.31) | 138.63 (13.97) | 139.13 (12.63)
Blood Pressure (diastolic) [Mean (Standard Deviation); unit: millimeters of mercury] | 73.34 (8.21) | 74.09 (9.37) | 73.71 (8.75)
Hemoglobin A1c [Mean (Standard Deviation); unit: mg/dL] | 7.72 (1.66) | 7.75 (1.56) | 7.73 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Number of PP-MI Sessions Completed by Participants
Description: Measured by number of PP-MI sessions completed by participants in the PP-MI group.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: sessions completed
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 35
sessions completed | 11 (4.45)

2. Secondary Outcome: Ease of PP Component
Description: Participants in the PP-MI group will provide ratings of ease after each PP exercise, measured on a 10-point Likert scale (0=very difficult; 10=very easy). Weekly ratings were averaged to provide an overall ease of the exercises.
Time Frame: Weeks 1-16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 35
units on a scale | 8.18 (1.98)

3. Secondary Outcome: Ease of MI Component
Description: Participants in the PP-MI group will provide ratings of ease after each MI exercise, measured on a 10-point Likert scale (0=very difficult; 10=very easy). Weekly ratings were averaged to provide an overall ease of the exercises.
Time Frame: Weeks 1-16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 35
units on a scale | 8.40 (1.83)

4. Secondary Outcome: Utility of PP Component
Description: Participants in the PP-MI group will provide ratings of utility after each PP exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 35
units on a scale | 8.78 (1.51)

5. Secondary Outcome: Utility of MI Component
Description: Participants in the PP-MI group will provide ratings of utility after each MI exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 35
units on a scale | 8.96 (1.40)

6. Secondary Outcome: Change in Moderate-Vigorous Physical Activity
Description: ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline, 16 weeks, and 24 weeks to assess the feasibility of doing so and to ensure adequate capture of physical activity.
Time Frame: Change from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants wore the Actigraph and provided adequate data at both follow-up time points.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 35 | 35
minutes/day
  16 weeks: number analyzed (Participants) | 25 | 27
  16 weeks | 3.88 (10.98) | -1.21 (9.76)
  24 weeks: number analyzed (Participants) | 22 | 23
  24 weeks | 2.75 (10.31) | 0.33 (12.09)

7. Secondary Outcome: Change in Physical Activity
Description: Measured by Actigraph accelerometer, in number of steps per day.
Time Frame: Change from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants wore the Actigraph and provided adequate data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 25 | 27
steps/day
  16 weeks | 904 (1206) | -379 (1228)
  24 weeks: number analyzed (Participants) | 22 | 23
  24 weeks | 222 (1410) | -290 (1301)

8. Secondary Outcome: Change in Sedentary Time
Description: Measured by Actigraph accelerometer, in minutes per day.
Time Frame: Change from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants wore the Actigraph and provided adequate data.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 25 | 27
minutes/day
  16 weeks | 19.68 (138.82) | 5.78 (74.75)
  24 weeks: number analyzed (Participants) | 22 | 23
  24 weeks | -11.84 (84.61) | 4.74 (79.95)

9. Secondary Outcome: Change in Positive Affect
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 16 and 24 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | 1.29 (5.68) | 0.41 (5.13)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 5.54 (6.09) | 4.21 (6.65)

10. Secondary Outcome: Change in Optimism
Description: Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change was calculated by subtracting the score at baseline from the score at 16 and 24 weeks. Higher scores indicate higher levels of optimism.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | 2.54 (4.38) | 0.55 (3.16)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 2.54 (3.79) | 0.43 (4.86)

11. Secondary Outcome: Change in Self-Efficacy for Exercise
Description: Measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assess self-efficacy barriers to exercise (Range: 0-90). Higher scores indicate higher efficacy expectations in relation to exercising. This was measured at Baseline, Week 16, and Week 24.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | 12.50 (22.66) | -9.55 (25.75)
  24 weeks: number analyzed (Participants) | 24 | 27
  24 weeks | 7.38 (21.97) | -7.81 (27.47)

12. Secondary Outcome: Change in Depression
Description: The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 16 and 24 weeks. Higher scores indicate higher levels of depression.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | -0.11 (3.19) | -0.72 (1.87)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 0.00 (3.02) | 0.46 (2.62)

13. Secondary Outcome: Change in Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 16 and 24 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | -1.04 (3.98) | -0.90 (2.23)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | -1.00 (3.44) | -0.96 (3.20)

14. Secondary Outcome: Change in Resilience
Description: Measured by the Brief Resilience Scale (BRS), a reliable scale which assesses a person's ability to recover from stress despite adversity (Range: 6-30). Higher scores indicate more resilience.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | -0.07 (3.95) | 0.00 (2.33)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | -0.25 (2.64) | 0.64 (2.33)

15. Secondary Outcome: Change in Perceived Social Support
Description: Measured by the Multidimensional Scale of Perceived Social Support (MSPSS), a scale that measures subjectively reported social support (Range: 12-84). Higher scores indicate more subjectively reported social support.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | -1.18 (19.88) | 3.83 (12.62)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 6.25 (14.86) | 5.57 (15.15)

16. Secondary Outcome: Change in Diabetes Self-Care
Description: Measured by the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more diabetes self-care activities.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed all follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | 0.79 (0.93) | 1.02 (1.03)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 0.97 (0.92) | 1.13 (1.20)

17. Other Pre Specified Outcome: Change in Medication Adherence
Description: Measured by Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum:100. Change was calculated by subtracting the score at baseline from the score at 16 weeks and 24 weeks. Higher scores indicate greater levels of medication adherence.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
percentage of medication taken
  16 weeks | 0.7 (5.4) | 0.3 (7.8)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 2.1 (4.1) | -0.4 (10.7)

18. Other Pre Specified Outcome: Change in Self-Reported Physical Activity
Description: Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. Change was calculated by subtracting the score at baseline from the score at 16 and 24 weeks.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed all follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: MET minutes per week
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 28
MET minutes per week
  16 weeks | 1512.41 (1957.69) | 96.10 (1704.43)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 912.72 (1096.29) | -87.80 (1585.93)

19. Other Pre Specified Outcome: Change in Physical Function
Description: Measured by the 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS), a well-validated measure of physical function that is highly responsive to changes in a patient's physical function status (Range: 20-100). Higher scores indicate better physical function.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 29
score on a scale
  16 weeks | 0.04 (5.72) | 0.31 (4.42)
  24 weeks: number analyzed (Participants) | 24 | 28
  24 weeks | 2.83 (4.67) | 0.96 (5.27)

20. Other Pre Specified Outcome: Change in Pain-Related Disability
Description: Measured by the Pain Disability Index (PDI), a well-validated measure of the extent to which pain interferes with different daily activities (Range 0-70). Higher scores indicate greater interference from pain.
Time Frame: Change in score from Baseline to 16 weeks, and Baseline to 24 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 28
score on a scale
  16 weeks | 1.11 (13.68) | -5.18 (10.50)
  24 weeks: number analyzed (Participants) | 24 | 27
  24 weeks | -2.83 (9.18) | -1.22 (13.65)

21. Other Pre Specified Outcome: Change in Weight
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 26
pounds | -2.08 (5.68) | 0.09 (4.88)

22. Other Pre Specified Outcome: Change in Body Mass Index (BMI)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 27 | 26
kg/m^2 | -0.28 (1.11) | 0.00 (0.73)

23. Other Pre Specified Outcome: Change in Blood Pressure (Systolic)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 27 | 25
millimeters of mercury | -5.52 (15.99) | -1.08 (17.21)

24. Other Pre Specified Outcome: Change in Blood Pressure (Diastolic)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 27 | 25
millimeters of mercury | -3.00 (7.76) | -0.36 (11.28)

25. Other Pre Specified Outcome: Change in Hemoglobin A1c
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
Number analyzed (Participants) | 28 | 26
mg/dL | 0.10 (1.09) | 0.10 (0.44)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events are "any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom or disease...whether or not associated with the subject's participation in the research."
Arm/Group | Positive Psychology + Motivational Interviewing | Diabetes Education
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 4/35 | 0/35
Other Adverse Events (participants affected / at risk) | 12/35 | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=35) | Diabetes Education (N=35)
Leg infection (Infections and infestations) | 1 (1) | 0 (0) — Participant reported having been hospitalized due to a leg infection.
Unexpected Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) — Two participants were hospitalized for atrial fibrillation.
Unexpected acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant was hospitalized for acute respiratory failure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=35) | Diabetes Education (N=35)
Unexpected hypoglycemia (Endocrine disorders) | 1 (1) | 2 (4) — One participant in the PP-MI group reported one episode of hypoglycemia; one participant in the Diabetes Education group reported one episode of hypoglycemia, and another participant in the Diabetes Education reported three episodes of hypoglycemia.
Cat bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant went to the ED because of a cat bite.
Unexpected abdominal pain and diarrhea (General disorders) | 0 (0) | 1 (1) — Participant went to an urgent care clinic due to abdominal pain and diarrhea.
Unexpected nose bleed (General disorders) | 0 (0) | 1 (1) — Participant went to the ED due to a nose bleed that lasted more than 30 minutes.
Unexpected ear fullness (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Participant went to the ED due to ear fullness.
Unexpected dizziness and abdominal pain (General disorders) | 0 (0) | 1 (1) — Participant went to the ED due to dizziness and abdominal pain.
Unexpected fall (General disorders) | 3 (5) | 0 (0) — Three participants reported falls. Two participants reported having experienced a fall while going about their daily activities, and one participant reported having experienced three separate falls while going about their daily activities.
Unexpected leg cramps (General disorders) | 2 (2) | 0 (0) — Two participants reported experiencing leg cramps while exercising.
Unexpected kidney stone (General disorders) | 1 (1) | 0 (0) — Participant went to the ED because of a kidney stone.
Unexpected flank pain (General disorders) | 1 (1) | 0 (0) — Participant went to the ED due to flank pain caused by recent kidney stone.
Unexpected gastrointestinal problems (Gastrointestinal disorders) | 0 (0) | 1 (1) — Participant reported having an upset stomach and loose stools after starting a new medication prescribed by their primary care physician.
Unexpected shortness of breath (General disorders) | 1 (1) | 0 (0) — Participant went to the ED due to shortness of breath.
Unexpected ankle injury (General disorders) | 1 (1) | 0 (0) — Participant reported having torn a ligament in their ankle.
Unexpected episode of high blood pressure (General disorders) | 1 (1) | 0 (0) — Participant went to the ED due to an episode of high blood pressure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT03164538/Prot_SAP_000.pdf